CLINICAL TRIAL: NCT00001208
Title: Botulinum Toxin for the Treatment of Neurological Disorders
Brief Title: Botulinum Toxin for the Treatment of Involuntary Movement Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 850195; 85-N-0195
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-11-07

CONDITIONS: Movement Disorders
Keywords: Botulinum Toxin; BTW; Natural History
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients 2 years and older, will be eligible for participation if they have a disorder that, in the judgment of the treating physician, might be amenable to treatment with BTX. Applicable disorders include but are not limited to dystonia, hemifacial spasm, blepharospasm, tremor, spasmodic dysphonia, tics, vocal fold tremor, oral lingual dyskinesia, tardive dyskinesia, spasticity, and spasmodic dysphonia.

SUMMARY:
BTX has been used since the 1980s in support of the research mission of NINDS. Initial studies were focused on expanding the applicability of BTX treatment to movement disorders and exploring new indications. We evaluated the efficacy of an alternative serotype, type F. Under other protocols, we continue to study the physiology of movement disorders and BTX response.

The application of BTX therapy to movement disorders requires an understanding of BTX preparation and handling. The treatment must be tailored to the disorder under treatment and to its expression in the individual patient. Users must know the specific techniques of injection, including the use of EMG and ultrasound guidance. This protocol allows us to train physicians in all aspects of the use of BTX. It also provides us with a cohort of patients, receiving a standard method of treatment and with a stable response to BTX injection, for participation in other protocols on movement disorders and on the responses to BTX injection.

DETAILED DESCRIPTION:
The efficacy of botulinum toxin (BTX) has now been demonstrated for a variety of diseases associated with involuntary muscles spasms or movement. The application of botulinum toxin therapy to movement disorders requires treatment tailored to the individual patient and specific techniques of injection. This protocol 1) allows us to follow the natural history of subjects with movement disorders who receive standard botox injections for treatment of movement disorders and 2) allows us to provide botulinum toxin injections for patients participating in other NIH studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients 2 years and older, will be eligible for participation if they have a disorder that, in the judgment of the treating physician, might be amenable to treatment with BTX.
  2. Applicable disorders include but are not limited to dystonia, hemifacial spasm, blepharospasm, tremor, spasmodic dysphonia, tics, vocal fold tremor, oral lingual dyskinesia, tardive dyskinesia, spasticity, and spasmodic dysphonia.

EXCLUSION CRITERIA:

1. Women who are planning on becoming pregnant, are pregnant or breastfeeding, for the duration of the condition.
2. Subjects who require treatment with an aminoglycoside antibiotic, until treatment is complete.
3. For laryngeal injections, subjects must have a paradoxical vocal fold movement with intermittent stridor due to either gastroesophageal reflux or emotional disorders

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a movement disorder will be enrolled.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1989-10-26 (Actual)

PRIMARY OUTCOMES:
Study Natural History- data analysis | Ongoing
  Data regarding the movement disorder of the subject and observations of their standard treatment will be collected. Data may be used for future research questions that are related to subjects movement disorder and/or treatment.
Maintain cohort of subjects | Ongoing
  To maintain a cohort of patients with dystonia and other movement disorders for participation in other studies on the physiology of dystonia and BTX injection

CONTACTS AND LOCATIONS:
Overall Officials: Debra J Ehrlich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD stored in the database will be shared. @@@@@@@@@@@@We may share identifiable research data with other NIH protocols, when subjects are co-enrolled. Data can be shared with other protocols, investigators, and subject health care and medical team upon subject requests and permissions. Data that may be shared are demographics, diagnosis, botulinum toxin injections (including site, dose, localication technique), response to injections, assessments from clinical evaluations and clinical rating scales or test results that are conducted for each subject. Data that is shared may be stripped of identifiers and may be coded ( de-identified ) or unlinked from an identifying code ( anonymized ). When coded data is shared, the key to the code will not be provided to collaborators, but will remain at NIH. @@@@@@@@@@@@
Supporting Information: Study Protocol
Time Frame: Data will be shared indefinitely.
Access Criteria: We do plan on broad data sharing. Therefore, there will be no restrictions on whom the data can be shared with.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1985-N-0195.html